CLINICAL TRIAL: NCT04256460
Title: Shanghai Community Prediabetes Standardized Management Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Collaborators: Shanghai Municipal Center for Disease Control and Prevention (Other)
Responsible Party: Principal Investigator, Weiping Jia, Professor, Director of Shanghai Diabetes Institute, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Shanghai6
Record Dates: First submitted 2019-10-16; First posted 2020-02-05 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: PreDiabetes
Keywords: prediabetes; life style intervention; peer support; self management support; primary healthcare; community
MeSH Terms: conditions — Prediabetic State | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Behavior intervention including health education on diet, exercises and self management support through peer support, and also receive regular care and follow up in community health centers
  Interventions: Behavioral: Healthy diet, regular exercises and peer support
- Control arm (No Intervention): Receiving regular care and follow up in Community health centers

INTERVENTIONS:
Behavioral: Healthy diet, regular exercises and peer support — After assessing the exercise and nutritional status of the participants, health staff in community health centers implemented personalized healthy diet and regular exercises intervention, including coaching on healthy exercises and developing personalized dietary prescriptions for participants. Besides, peer support is implemented as a self management strategy in community health service centers or community self management groups to enhance the behavioral change support for these participants.
  Arms: Intervention arm

SUMMARY:
Participants with prediabetes is the key targets for diabetes prevention. So, in order to further strengthen and standardize the management of participants with prediabetes in the communities, the investigators start this project of standardized management of participants with prediabetes in communities of Shanghai. Explore the standardized management model for prediabetes participants within primary healthcare settings in Shanghai, to reduce the risk factors of diabetes, improve the blood glucose control, and the quality of life of participants with prediabetes.

DETAILED DESCRIPTION:
Participants with prediabetes is the key targets for diabetes prevention. So, in order to further strengthen and standardize the management of participants with prediabetes in the communities, the investigators start this project of standardized management of participants with prediabetes in communities of Shanghai. Explore the standardized management model for prediabetes participants within primary healthcare settings in Shanghai, to reduce the risk factors of diabetes, improve the blood glucose control, and the quality of life of participants with prediabetes.

Through the collaboration the Shanghai Municipal Center for Disease Control & Prevention network, this investigators will implement prediabetes screening and lifestyle intervention in around 50 community health service centers in Shanghai. Life-style interventions including exercise and diet, and diabetes prevention knowledge will be integrated into "train-the-trainers" workshops. Trainings will be provided to community health service staff and peer supporters or social workers.

ELIGIBILITY:
Inclusion Criteria:

* Chinese residents
* Adult age ≥ 18 years old, 35-75 years old preferred
* Participants receiving prediabetes management of the basic public health services package in community health centers
* BMI≥24 kg/m2 or central obesity (Waist circumference≥90 cm in males，Waist circumference≥85 cm in females) or Hypertension (SBP≥140 mmHg and/or DBP≥90 mmHg) preferred
* Signed informed consents and willing to participate

Exclusion Criteria:

* With serious chronic diseases, tumors, acute and chronic infectious diseases, limb movement disorders, and any mental illnesses
* Women during pregnancy or breastfeeding
* With excessive drinking or illicit drug use
* Unwilling to participate in the project
* Histories of severe cardiovascular events (myocardial infarction, stroke, acute coronary syndrome, or transient ischemic attack (TIA))

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change of BMI from baseline at 12 months | Baseline, 12 months
  body mass index, using the examination results of height (cm) and weight (kg)

SECONDARY OUTCOMES:
Change of HbA1c from baseline at 12 months | Baseline, 12 months
  hemoglobin A1c (%)
Change of Waist circumference from baseline at 12 months | Baseline, 12 months
  Waist circumference (cm)
Change of Fasting Plasma Glucose from baseline at 12 months | Baseline, 12 months
  fasting plasma glucose (mmol/L)
Change of Blood Pressure from baseline at 12 months | Baseline, 12 months
  Blood pressure including systolic blood pressure and diastolic blood pressure (mmHg)
Change of Total Cholesterol from baseline at 12 months | Baseline, 12 months
  total cholesterol (mmol/L)
Change of Triglyceride from baseline at 12 months | Baseline, 12 months
  Triglyceride (mmol/L)
Change of High density lipoprotein cholesterol from baseline at 12 months | Baseline, 12 months
  High density lipoprotein-Cholesterol (mmol/L)
Change of Low density lipoprotein cholesterol from baseline at 12 months | Baseline, 12 months
  Low density lipoprotein-Cholesterol (mmol/L)

OTHER OUTCOMES:
Change of Liver Functioning from baseline at 12 months | Baseline, 12 months
  alanine transaminase (U/L), Aspartate transaminase (U/L), Alkaline phosphatase (U/L), glutamyltransferase (U/L)
Change of Urine Albumin/Creatinine Ratio from baseline at 12 months | Baseline, 12 months
  Albumin (mg/L), Creatinine (mmol/L)
Change of Bilirubin from baseline at 12 months | Baseline, 12 months
  Total bilirubin (μmol/L), Direct bilirubin (μmol/L)
  Total bilirubin (μmol/L), Direct bilirubin (μmol/L)
Change of Blood Urea from baseline at 12 months | Baseline, 12 months
  Blood urea (mmol/L)
Change of Serum Creatinine from baseline at 12 months | Baseline, 12 months
  Serum creatinine (μmol/L)
Change of Uric Acid from baseline at 12 months | Baseline, 12 months
  Uric acid (μmol/L)
Change of oral glucose tolerance test-2 hour from baseline at 12 months | Baseline, 12 months
  oral glucose tolerance test-2 hour (mmol/L)
Change of Diabetes Self Care Behaviors from baseline at 12 months | Baseline, 12 months
  9 items from Summary of Diabetes Self Care Activities and Behavioral Risk Factor Surveillance System. Items 1-7 measure diabetes self care activities during the previous 7 days. Items 1, 2, 4-7 are assessed on a scale of 0 to 7 days. Item 3 is assessed on scale of 1-4, where 1 represents very low levels of daily activity and 4 represents very high levels of daily activity. Items 8 and 9 are yes/no questions that measure cigarette intake over the past 7 and 30 days.
Change of General Quality of Life from baseline at 12 months | Baseline, 12 months
  6-item Euro quality-of-life-5D, a standardized instrument for measuring generic health status. The respondents are asked to choose one of the statements which best describes their health status on the surveyed day. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). Item 6 is the visual analogue scale, in which respondents are asked to mark their health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100, where 0 corresponds to "the worst health you can imagine", and 100 corresponds to "the best health you can imagine"
Change of Diabetes Quality of Life from baseline at 12 months | Baseline, 12 months
  4-item Diabetes Distress Scale, an abbreviated version of the 17-item Diabetes Distress Scale. The respondents are asked to respond to which degree each of the items has bothered them in the past month on a 6-point scale (1-6), where 1 is not a brother and 6 is very bothersome. Scores are summed and divided by 4 to calculate the mean. Mean scores of 3 or higher (moderate distress) are considered worthy of clinical attention.
Change of Depression from baseline at 12 months | Baseline, 12 months
  8-item Patient Health Questionnaire (PHQ), the PHQ-9 minus the last question on suicidal thoughts. The PHQ is a standard instrument used in primary care settings to screen for the presence and severity of depression. The respondents are asked how often they have been bothered by each of the 8 items in the past 2 weeks on a 4 point scale (0-3), where 0 is "not all" and 3 is "nearly every day". The scores for each item are summed to produce a total score between 0 and 24 points. A total score of 0 to 4 represents no significant depressive symptoms. A total score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe.
Change of Insulin Attitudes from baseline at 12 months | Baseline, 12 months
  6 questions
Change of Neighborhood Interactions from baseline at 12 months | Baseline, 12 months
  6 questions
Change of Peer Support Engagement and Health Care Utilization from baseline at 12 months | Baseline, 12 months
  5 questions
Change of General information and risk factors questionnaire from baseline at 12 months | Baseline, 12 months
  Demographic questions, medical histories, risk factors including family history, smoking, alcohol drinking, diet, and exercises, medication information and adherence.
Change of C-reaction protein from baseline at 12 months | Baseline, 12 months
  C-reaction protein

CONTACTS AND LOCATIONS:
Locations (53):
- China (53):
  - Anting community health service center, Shanghai, Shanghai Municipality
  - Baihe community health service center, Shanghai, Shanghai Municipality
  - Beiwaitan community health service center, Shanghai, Shanghai Municipality
  - Caoyang community health service center, Shanghai, Shanghai Municipality
  - Changfeng baiyu community health service center, Shanghai, Shanghai Municipality
  - Changfeng changfeng community health service center, Shanghai, Shanghai Municipality
  - Changqiao community health service center, Shanghai, Shanghai Municipality
  - Changshou community health service center, Shanghai, Shanghai Municipality
  - Changzhengzhen community health service center, Shanghai, Shanghai Municipality
  - Chendun community health service center, Shanghai, Shanghai Municipality
  - Chonggu community health service center, Shanghai, Shanghai Municipality
  - Dahua community health service center, Shanghai, Shanghai Municipality
  - Dongjing community health service center, Shanghai, Shanghai Municipality
  - Fangsong community health service center, Shanghai, Shanghai Municipality
  - Fenglin community health service center, Shanghai, Shanghai Municipality
  - Ganquan community health service center, Shanghai, Shanghai Municipality
  - Hongmei community health service center, Shanghai, Shanghai Municipality
  - Huamu community health service center, Shanghai, Shanghai Municipality
  - Huangdu community health service center, Shanghai, Shanghai Municipality
  - Huinan community health service center, Shanghai, Shanghai Municipality
  - Jiangwan community health service center, Shanghai, Shanghai Municipality
  - Jinqiao community health service center, Shanghai, Shanghai Municipality
  - Jinyang community health service center, Shanghai, Shanghai Municipality
  - Juyuanxinqu community health service center, Shanghai, Shanghai Municipality
  - Kangjian community health service center, Shanghai, Shanghai Municipality
  - Liantang community health service center, Shanghai, Shanghai Municipality
  - Longhua community health service center, Shanghai, Shanghai Municipality
  - Luodian community health service center, Shanghai, Shanghai Municipality
  - Luojing community health service center, Shanghai, Shanghai Municipality
  - Malu community health service center, Shanghai, Shanghai Municipality
  - Miaohang community health service center, Shanghai, Shanghai Municipality
  - Nanjingxi Road community health service center, Shanghai, Shanghai Municipality
  - Nanxiang community health service center, Shanghai, Shanghai Municipality
  - Nicheng community health service center, Shanghai, Shanghai Municipality
  - Puxing community health service center, Shanghai, Shanghai Municipality
  - Qilian community health service center, Shanghai, Shanghai Municipality
  - Quyang community health service center, Shanghai, Shanghai Municipality
  - Sheshan community health service center, Shanghai, Shanghai Municipality
  - Shiquan community health service center, Shanghai, Shanghai Municipality
  - Songnan community health service center, Shanghai, Shanghai Municipality
  - Tangzhen community health service center, Shanghai, Shanghai Municipality
  - Taopuzhen community health service center, Shanghai, Shanghai Municipality
  - Taopuzhen No.2 community health service center, Shanghai, Shanghai Municipality
  - Tianlin community health service center, Shanghai, Shanghai Municipality
  - Waigang community health service center, Shanghai, Shanghai Municipality
  - Xianghuaqiao community health service center, Shanghai, Shanghai Municipality
  - Xiaokunshan community health service center, Shanghai, Shanghai Municipality
  - Yichuan community health service center, Shanghai, Shanghai Municipality
  - Yuepu community health service center, Shanghai, Shanghai Municipality
  - Zhaoxiang community health service center, Shanghai, Shanghai Municipality
  - Zhenruzhen community health service center, Shanghai, Shanghai Municipality
  - Zhongshan community health service center, Shanghai, Shanghai Municipality
  - Zhujiajiao community health service center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No